CLINICAL TRIAL: NCT03277521
Title: Intermittent Theta Burst Stimulation to Promote Motor Re-education After Upper Limb Reconstruction in Tetraplegia
Brief Title: Theta Burst Stimulation to Promote Motor Re-education in Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Medical University of South Carolina (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20010643; FP00005482 (Other: Virginia Commonwealth University); P2CHD086844 (NIH)
Record Dates: First submitted 2017-08-24; First posted 2017-09-11 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Quadriplegia/Tetraplegia
MeSH Terms: conditions — Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neurologically Normal (Active Comparator): Neurologically normal subjects (i.e., nonimpaired) will be recruited for participation in three sessions of intermittent theta burst stimulation (iTBS), each consisting of sham iTBS applied to the hotspot of the target muscle and active iTBS; sham iTBS always be will administered first to minimize the potential for carry over effects. Sessions will be separated by at least 3 days to minimize the potential for carry over effects. Before and 10, 20 and 30 minutes after each iTBS session, motor evoked potentials (MEPs) will be recorded in order to quantify changes in corticomotor excitability.
  Interventions: Other: Intermittent theta burst stimulation
- Quadriplegia (Active Comparator): Individuals with quadriplegia will be recruited for participation in three sessions of intermittent theta burst stimulation (iTBS), each consisting of sham iTBS applied to the hotspot of the target muscle and active iTBS; sham iTBS always be will administered first to minimize the potential for carry over effects. Sessions will be separated by at least 3 days to minimize the potential for carry over effects. Before and 10, 20 and 30 minutes after each iTBS session, motor evoked potentials (MEPs) will be recorded in order to quantify changes in corticomotor excitability.
  Interventions: Other: Intermittent theta burst stimulation
- Quadriplegia with upper limb reconstruction (Active Comparator): Individuals with quadriplegia and upper limb reconstruction will be recruited for participation in three sessions of intermittent theta burst stimulation (iTBS), each consisting of sham iTBS applied to the hotspot of the target muscle and active iTBS; sham iTBS always be will administered first to minimize the potential for carry over effects. Sessions will be separated by at least 3 days to minimize the potential for carry over effects. Before and 10, 20 and 30 minutes after each iTBS session, motor evoked potentials (MEPs) will be recorded in order to quantify changes in corticomotor excitability.
  Interventions: Other: Intermittent theta burst stimulation

INTERVENTIONS:
Other: Intermittent theta burst stimulation — Intermittent theta burst stimulation (iTBS) is a non-invasive brain stimulation technique that can increase corticomotor excitability.

SUMMARY:
A repetitive, non-invasive brain stimulation technique referred to as theta burst stimulation can modulate corticomotor excitability and therefore has great rehabilitative potential for individuals with neurologic deficits, including individuals with spinal cord injury (SCI). In particular, intermittent theta burst stimulation (iTBS) can increase corticomotor excitability and may be a useful adjunct to physical rehabilitation to promote motor re-education after upper limb reconstruction in individuals with tetraplegia. Upper limb reconstruction involves surgical transfer of a non-paralyzed tendon or nerve with a redundant or less important function to perform a more critical function. Upper limb reconstruction is intended to help individuals achieve their goals related to activities of daily living and independence in the community. Outcomes after reconstruction are variable and depend largely on the efficacy of motor re-education of the transferred muscle to perform a new function. The long-term goal of our research is to determine whether iTBS combined with physical rehabilitation can improve motor re-education after reconstruction. As a first step, the purpose of this proposal is to determine the effect of iTBS on corticomotor excitability of proximal muscles in nonimpaired individuals and two groups of individuals with tetraplegia: individuals with and without upper limb reconstruction.

ELIGIBILITY:
Inclusion Criteria for all subjects with tetraplegia:

* Injury to the lower cervical spinal cord at least one year prior to the date of participation
* Motor function classified according to the American Spinal Injury Association International Standards for Neurological Classification of Spinal Cord Injury at levels ranging from C5-C8

Inclusion criteria for the subjects with tetraplegia and upper limb reconstruction:

• At least one year post-operative from tendon or nerve transfer surgery of the upper limb

Exclusion criteria for all subjects with tetraplegia:

* Presence of concurrent severe medical illness, including unhealed decubiti, use of baclofen pumps, existing infection, cardiovascular disease, significant osteoporosis, or a history of pulmonary complications.
* Metal implant near head or neck
* Risk of seizure of history of seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Change in corticomotor excitability | Each subject will participate in five sessions, each session separated by 3 days. After each session, changes in corticomotor excitability will be measured. Changes in excitability will be reported through study completion, an average of one month.
  Corticomotor excitability will be measured via motor evoked potential amplitudes in response to transcranial magnetic stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Carrie L Peterson, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mittal N, Majdic BC, Peterson CL. Intermittent theta burst stimulation modulates biceps brachii corticomotor excitability in individuals with tetraplegia. J Neuroeng Rehabil. 2022 Jul 17;19(1):73. doi: 10.1186/s12984-022-01049-9. PMID 35843943

DOCUMENTS (1):
  • Informed Consent Form (2019-08-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT03277521/ICF_000.pdf